CLINICAL TRIAL: NCT05675839
Title: THE EFFECT OF PROFESSIONAL FILMS ON PROFESSIONAL PRIDE IN NURSING STUDENTS-Randomized Controlled Study
Brief Title: Professional Pride in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Cevriye Ozdemir, Asst.Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BSAKN1D055
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Professional Role
MeSH Terms: interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: This study were conducted between September and December 2022 on 102 volunteer students studying in the Department of Nursing in Turkey. The inclusion criteria were as follows being 18 years old or over, being a firs year student, be in the classroom on training day. The students included in the study were randomly divided into two groups.Experimental group watched a documantary and a movie about nursing profession and Control group had no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Before the intervention, students filled the "Nursing Professional Pride Scale". Nursing students watched a documentary and a movie about nursing profession. After the intervention, students filled the "Nursing Professional Pride Scale".
  Interventions: Other: Film (Wit) and a documentary (First Turkish Nurse-Safiye Hüseyin Elbi's Life)
- Control (No Intervention): First of all, Control group filled the "Nursing Professional Pride Scale". The control group have no intervention. They filled the scale again, after 2 week.

INTERVENTIONS:
Other: Film (Wit) and a documentary (First Turkish Nurse-Safiye Hüseyin Elbi's Life) — Film (Wit) (https://www.youtube.com/watch?v=2s4ozvI_hzY&t=160s) and a documentary (First Turkish Nurse-Safiye Hüseyin Elbi's Life) (https://www.youtube.com/watch?v=XsabHOiF0CY&t=284s)
  Arms: Experimental

SUMMARY:
Nursing is a scientific discipline based on professional values, principles and standards. Nursing care is a holistic and continuous approach. Therefore, nurses spend more time interacting with patients or healthy individuals than other healthcare professionals. Effective and quality nursing care depends on professional attitudes, perceptions and satisfaction. Movies are recognized as effective educational resources to encourage the retention of knowledge and the development of desired behaviors. Therefore, in this study, it is aimed to determine the effect of movies about the profession on the professional pride of nursing students.

DETAILED DESCRIPTION:
The study was conducted to determine the effect of professional films on the professional pride of nursing students.

The study is a single-center, randomized controlled experimental study. The study, which was conducted in randomized controlled experimental design, included 102 students enrolled in the first year of nursing faculty of a state university in the 2022-2023 academic year.

Sampling Inclusion Criteria: Individuals over the age of 18, who agreed to participate in the study in written and verbal form, and participated in all phases of the study were included.

The students were randomly divided into two groups, 66 experimental and 66 control groups. Since there were students who did not complete the study in both groups, the study was completed with a total of 102 students, 57 of which were experimental and 45 were control.

Data were collect with "Sociodemographic Data Form" and "Nursing Professional Pride Scale" .

Written permission were obtained from the individuals who volunteered to participate in the study, and "Sociodemographic Data Form" and "Nursing Professional Pride Scale" were applied to all students.

The names of all students were written in alphabetical order, and students were divided into "Experimental" or "Control" groups using the random numbers table.

Intervention in Experimental Group:First of all, movie or documentary suggestions on the professional role of nursing, available on YouTube, were received from 5 nurse academicians who are experts in the field of Nursing Fundamentals. A film (Wit (2001), and a documentary (The First Turkish Nurse- Safiye Huseyin Elbi's Life) were selected by the researchers with agreed. The students in the experimental group were asked to watch a documentary and then a movie with a one-week break. After the interventions "Nursing Professional Pride Scale" were applied to intervention groups.

Intervention in Control Group: No intervention. After two weeks "Nursing Professional Pride Scale" were applied to control groups.

In the analysis of the data, nominal variables were evaluated as frequency and percentage, and ordinal variables were evaluated as mean and standard deviation. Chi-square relationship between scales, Spearman's rho, Mann-Whitney U Test and Wilcoxon Signad Rank Test were used.

ELIGIBILITY:
Inclusion Criteria:

* Over18 years old
* Being 1st year student
* who agreed to participate in the study in written and verbal form,
* participated in all phases of the study were included

Exclusion Criteria:

-Not being volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Data of the students | Baseline
  The form in which the socio-demographic data of the students such as age and gender are questioned.
Nursing Professional Pride Scale | Baseline and 2 week later.
  The Turkish version of the Nursing Professional Pride Scale (NPPS-TR) were used. The Nursing Professional Pride Scale (NPPS) was developed by JaeHee et al. to measure levels of professional pride in nurses. The scale consists of 27 items and five subscales. The items are scored on a five-point Likert-type scale of (1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree). The subscales are feeling of vocation, (six items, 1, 2, 3, 4, 5, and 6), role satisfaction (six items, 7, 8, 9, 10, 11, and 12), role of problem solver (six items, 13, 14, 15, 16, 17, and 18), self-achievement (four items, 19, 20, 21, and 22), and willingness to stay (five items, 23, 24, 25, 26, and 27). The total score ranges from 27 to 135, with higher scores indicating greater professional pride.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Kabuk, PhD, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If it is necessary for the ethical issue, investigators can share.

REFERENCES:
- [Result] Aydin A, Erbas A, Kaya Y. Nursing Professional Pride Scale: Turkish adaptation and psychometric properties. Perspect Psychiatr Care. 2022 Jan;58(1):206-213. doi: 10.1111/ppc.12812. Epub 2021 Apr 24. PMID 33896028
- [Result] Jeon J, Lee E, Kim E. [Development of an Instrument to Assess the Nursing Professional Pride]. J Korean Acad Nurs. 2020 Apr;50(2):228-241. doi: 10.4040/jkan.2020.50.2.228. Korean. PMID 32376811
- See also: First Turkish Nurse-Safiye Hüseyin Elbi's Life (Documentary) — http://www.youtube.com/watch?v=XsabHOiF0CY&t=284s
- See also: Wit (Film) — http://www.youtube.com/watch?v=2s4ozvI_hzY&t=160s